CLINICAL TRIAL: NCT02751684
Title: EUROpE RSI-Study (EURopean Online Evaluation) - Pan-european Online-survey About Rapid Sequence Induction (RSI) by Anesthetists
Brief Title: EUROpE-RSI (EURopean Online Evaluation RSI Study)
Acronym: EUROpE-RSI
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Köln (Other)
Responsible Party: Sponsor
Other Study IDs: UKoln
Record Dates: First submitted 2016-04-11; First posted 2016-04-26 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Rapid Sequence Induction
Keywords: Rapid Sequence Induction; European; Evaluation; EUROpE RSI; Standards; RSI

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators want to identify and show differences in standards and procedures of in-hospital rapid sequence induction by collecting data with an online survey for anaesthetist in Europe.

DETAILED DESCRIPTION:
The study is designed as a web-based online survey for anaesthetist in Europe. They will be invited via mail, as members of the European Society of Anaesthesiology (ESA), the participation is voluntary.

The survey contains 30 items about the standards and procedures of in-hospital rapid sequence induction (RSI). There will be a selection of possible answers, only a few items contains free-text answers.

The study collects only personal data to age, country, gender and level of training.

The collected data should identify differences in the procedures of RSI.

ELIGIBILITY:
Inclusion Criteria:

* Emergency physician

Exclusion Criteria:

* None Emergency physician

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Emergency physicians from europe; e.g. members of the European Society of Anaestesiology
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Differences in the procedure of the RSI (Rapid sequence induction) | 04.30.2016-10.30.2016
  The questionnaire date will be collected up to 6 month and processed with Microsoft Excel.

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital of Cologne, Cologne, North Rhine-Westphalia, Germany